CLINICAL TRIAL: NCT01403155
Title: PHASE I, OPEN-LABEL, SAFETY, TOLERABILITY, AND IMMUNOGENICITY STUDY OF AN H5 INFLUENZA PLASMID VACCINE (INO-3401) IN HEALTHY ADULTS PREVIOUSLY VACCINATED WITH VGX-3400X
Brief Title: A Follow-On Study With an H5 Influenza Vaccine for Subjects Who Participated in Study FLU-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLU-002
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: H5N1; Avian Influenza; DNA Vaccine; Intradermal (ID) Injection; Electroporation; Healthy Adults
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will receive 0.9mg/mL of study vaccine (INO-3401 DNA plasmid vaccine) at Day o and Month 3.
  Interventions: Biological: INO-3401 + EP

INTERVENTIONS:
Biological: INO-3401 + EP — All subjects will receive 0.9mg/mL of study vaccine (INO-3401 DNA plasmid vaccine)at Day 0 and Month 3.

SUMMARY:
DNA vaccines consist of small pieces of DNA also known as plasmids, and have several potential advantages over traditional vaccines. Thus far, DNA vaccines appear to be well tolerated in humans. The investigators have developed a DNA vaccine, INO-3401, which includes plasmids targeting the proteins of the H5N1 avian influenza virus. The vaccine will be delivered via electroporation (EP) which uses the CELLECTRA constant current device to deliver a small electric charge following injection, since animal studies have shown that this delivery method increases the immune response to vaccine. The vaccine will be given to up 30 healthy adult subjects who have participated in study FLU-001. It is hypothesized that a booster dose with INO-3401 + EP will be well tolerated and immunogenic.

DETAILED DESCRIPTION:
The use of DNA plasmids containing genes that express viral antigens may be a promising way to formulate a vaccine that can effectively prevent infection and disease caused by the H5N1 avian influenza virus. Plasmid vectors are simple to construct and are easy to manufacture at a relatively low cost. Vaccination with plasmids that express influenza proteins should induce the development of serum antibodies and might also induce significant quantities of secretory IgA antibodies and/or CMI. The DNA sequences included in the vaccine could also result in the proliferation of T lymphocytes that could broaden the effectiveness of the vaccine to include variant strains of H5N1 with antigenically modified HA (i.e., drifted strains).

Electroporation (EP) is a technology in which a transmembrane electrical field is applied to increase the permeability of cell membranes to create microscopic pathways (pores) and thereby enhance the uptake of drugs, vaccines, or other agents into target cells. Their presence allows macromolecules, ions, and water to pass from one side of the membrane to the other. The presence of a constant field influences the kinetics of directional translocation of the macromolecular plasmid, such that the plasmid delivery in vivo has been sufficient to achieve physiological levels of secreted proteins. Intradermal (ID) injection of plasmid followed by EP has been used very successfully to deliver therapeutic genes that encode for a variety of hormones, cytokines, or enzymes in a variety of species. EP is currently being used in humans to deliver cancer vaccines and therapeutics as well as in gene therapy. The expression levels are increased by as much as 3 orders of magnitude over plasmid injection alone.

The use of EP via the CELLECTRA® device should increase the expression of H5N1 influenza virus genes in the INO-3401 DNA vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines. If required by local law, candidates must also authorize the release and use of protected health information (PHI);
* Enrollment in and received at least one vaccination in study FLU-001;
* Adults of either gender 18-50 years of age at entry;
* Healthy subjects as judged by the Investigator based on medical history, physical examination, and negative pregnancy test for Women of child-bearing potential (WOCBP) prior to enrollment and administration of study drug;
* Current nonsmoker;
* WOCBP agree to remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc), or have a partner who is sterile (i.e.,vasectomy) through Month 4 of the study;
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Subjects with grade 3 or 4 CPK elevation;
* Pregnant or breastfeeding subjects;
* Any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site (excluding inhaled and eye drop-containing corticosteroids) or the use of other immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study vaccine administration;
* Administration of any blood product within 3 months of enrollment;
* Prior receipt of an H5N1 influenza vaccine at any time;
* Subjects with a contraindications to influenza vaccination other than egg allergy (such as a history of Guillain-Barre Syndrome after receiving influenza vaccine);
* Administration of any vaccine other than VGX-3400X within 6 weeks of enrollment;
* Subject is currently participating or has participated in a study with an investigational compound other than FLU-001 within 30 days of signing informed consent;
* Subjects with cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);
* Subjects with a history of seizures (unless seizure free for 5 years);
* Subjects with tattoos, scars, or active lesions/rashes within 2 cm of the site of vaccination/EP;
* Subjects with any implantable leads;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
* Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety | Day 0 through Month 9
  Frequency and severity of local and systemic reactogenicity, signs and symptoms, adverse events and serious adverse events.

SECONDARY OUTCOMES:
Humoral and cellular immune responses | Day 0 through Month 9
  Magnitude and frequency of antibody and cell-mediated immune responses to influenza proteins.
Tolerability | Day 0 and Month 3
  Tolerability by Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bagarazzi, MD, Study Director — Inovio Pharmaceuticals
Locations (2):
- United States (2):
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Accelovance, Rockville, Maryland

REFERENCES:
- See also: Sponsor's Website — http://www.inovio.com